CLINICAL TRIAL: NCT00748800
Title: An Affect Management Intervention for Juvenile Offenders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Larry K. Brown, M.D./Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21DA019245 (NIH)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: HIV prevention; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Affect Management
- 2 (Active Comparator)
  Interventions: Behavioral: General Health Promotion

INTERVENTIONS:
Behavioral: Affect Management — 5 session group intervention that focused on teaching affect management skills and included HIV prevention and sexual health training
  Arms: 1
Behavioral: General Health Promotion — 5 session group focused on delivering general health promotion information in didactic format
  Arms: 2

SUMMARY:
Adolescents are at risk for HIV because of sexual and drug behavior initiated during this developmental period. Adolescents in the juvenile justice system are at increased risk for HIV due to higher rates of substance use and psychopathology than their non-offending peers. Juvenile justice youth may therefore also be less likely to benefit from frequently used skills based interventions. It appears that emotional lability, frequently found in this population, disrupts skills learned. This project will implement and evaluate an affect management HIV prevention intervention for adolescents in a juvenile drug court program. Affect management and general health promotion interventions will be compared to determine which intervention best reduces risk behavior among adolescents in the drug court.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents enrolled in the juvenile drug court program

Exclusion Criteria:

* Adolescent is HIV positive
* Adolescent is pregnant
* Adolescent is developmentally delayed
* Adolescent has history of sexual crime

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2004-09; Primary Completion 2007-05 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Adolescent-reported sexual activity and condom use | 3 month post-intervention

SECONDARY OUTCOMES:
Adolescent substance use (self-report and urine toxicology screen results) | 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States